CLINICAL TRIAL: NCT06418113
Title: Neoadjuvant Radio-chemotherapy Safety Pilot Study in Patients With Glioblastoma
Acronym: GLINERA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Asociación de Afectados Por Tumores Cerebrales en España (ASATE) (Unknown)
Responsible Party: Principal Investigator, Juan Antonio Barcia Albacar, Professor, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/399
Record Dates: First submitted 2024-04-03; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma, IDH-wildtype; Radiotherapy; Complications; Cancer Brain
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Stereotactic biopsy will be performed on patients in the experimental group, who will then be discharged. If the histopathological diagnosis is not wildtype IDH non-mutated glioblastoma, the patient will be withdrawn from the study and receive conventional treatment. If wildtype IDH non-mutated glioblastoma is diagnosed, ten days after the biopsy, patients will undergo conformal hypofractionated stereotactic radiotherapy to the FLAIR hyperintense signal, including the contrast-enhancing tumor on T1, with a total dose of 3990 cGy at the margin in 15 fractions of 266 cGy, one session per day, five days a week, and concurrent temozolomide (TMZ) at 75 mg/m2/day for 7 days/week during the irradiation period (GEINO, 2016). Five weeks later, patients will undergo supramarginal resection guided by 5-ALA under intraoperative neurophysiological monitoring. Starting from 4 weeks post-surgery, TMZ will be administered for 6 months according to the Stupp protocol.
  Interventions: Radiation: hypofractionated stereotactic radiotherapy; Procedure: Stereotactic biopsy; Procedure: resection; Drug: Chemotherapy
- Stupp Protocol (Other): The Stupp protocol is a standard treatment regimen for glioblastoma, which involves a combination of radiotherapy and chemotherapy.
  Interventions: Procedure: resection; Radiation: radiotherapy Stupp protocol; Drug: Chemotherapy Stupp Protocol

INTERVENTIONS:
Radiation: hypofractionated stereotactic radiotherapy — conformal hypofractionated stereotactic radiotherapy to the FLAIR hyperintense signal, including the contrast-enhancing tumor on T1, with a total dose of 3990 cGy at the margin in 15 fractions of 266 cGy, one session per day, five days a week, and concurrent temozolomide (TMZ) at 75 mg/m2/day for 7 days/week during the irradiation period
  Arms: Experimental
Procedure: Stereotactic biopsy — Stereotactic biopsy
  Arms: Experimental
Procedure: resection — supramarginal resection guided by 5-ALA under intraoperative neurophysiological monitoring
Drug: Chemotherapy — 4 weeks post-surgery, temozolomide (TMZ) will be administered for 6 months
  Arms: Experimental
Radiation: radiotherapy Stupp protocol — radiotherapy + TMZ concurrently after 4 weeks of resection surgery, as per usual protocol: Three-dimensional radiotherapy planning to deliver a total dose of 60 Gy, with a fractionation of 2 Gy/day, 5 days/week, encompassing a 1-2 cm margin around the contrast-enhancing region defined on T1 imaging or the entire abnormal volume defined on T2 or FLAIR imaging (Li et al., 2016) + TMZ at 75 mg/m2/day for 7 days/week, for 6 weeks during radiotherapy.
  Arms: Stupp Protocol
Drug: Chemotherapy Stupp Protocol — temozolomide (TMZ) will be administered for 6 months according to the Stupp protocol.
  Arms: Stupp Protocol

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of neoadjuvant radiochemotherapy in the surgical resection of glioblastoma (GBM). The main questions it aims to answer are:

* What is the safety profile of neoadjuvant radiochemotherapy in terms of neurological deficit, radionecrosis, edema, headache, wound dehiscence, infection, and cerebrospinal fluid fistula?
* What is the efficacy of neoadjuvant radiochemotherapy in terms of progression-free survival, overall survival, cognitive function, and quality of life?

Participants will undergo the following tasks and treatments:

* Stereotactic biopsy and diagnosis confirmation.
* Conformal hypofractionated stereotactic radiotherapy with concurrent temozolomide.
* Supramarginal resection guided by 5-ALA under intraoperative neurophysiological monitoring.
* Maintenance temozolomide administration for 6 months.

Researchers will compare the group receiving neoadjuvant radiochemotherapy to the control group following the standard Stupp protocol to assess safety and efficacy outcomes.

DETAILED DESCRIPTION:
Objectives: To study the safety (primary) and efficacy (secondary) of neoadjuvant radiochemotherapy in the surgical resection of glioblastoma (GBM). Safety measures include: neurological deficit, radionecrosis (radiological and clinical), edema, headache, wound dehiscence, infection, and cerebrospinal fluid fistula. Efficacy measures include progression-free survival (PFS), overall survival (OS), cognitive function (MoCA Scale), and quality of life (EuroQol scales, EORTC QLQ-HN35, FACT-Br, and TWiST). Methods: Pilot safety and efficacy study in 6 patients compared to 6 controls. 2-year follow-up. A data safety monitoring committee will review the data one month after surgery for each of the first three patients to decide whether to stop or continue the study. Stereotactic biopsy will be performed, and if GBM is diagnosed, patients will undergo conformal hypofractionated stereotactic radiotherapy to the FLAIR hyperintense signal including the contrast-enhancing tumor on T1, with a total dose of 3990 cGy at the margin in 15 fractions of 266 cGy and concurrent temozolomide (TMZ). 5 weeks later, patients will undergo supramarginal resection guided by 5-ALA under intraoperative neurophysiological monitoring. 7 days after surgery, maintenance TMZ will be administered for 6 months. The control group will follow standard treatment (Stupp protocol). Data analysis will be performed using non-parametric tests. Samples from successive surgeries will be studied with histology, molecular biology, and cell cultures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Unifocal disease.
* Unilobar tumor.
* Clinical-radiological diagnosis of supratentorial unicentric high-grade glioma, eligible for macroscopically complete resection.

Exclusion Criteria:

* Multilobar tumor, interhemispheric or infratentorial extension, or multifocal disease.
* Midline shift greater than 1 cm.
* Intracranial hypertension symptoms requiring corticosteroid treatment.
* Synchronous neoplasia.
* Any contraindication for surgery, radiotherapy, or TMZ treatment.
* Cognitive impairment.
* Rejection of informed consent.
* Inability to follow up for 2 years.
* Women of childbearing potential according to the Clinical Trial Facilitation Group (CTFG) criteria. (https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2020_09_HMA_CTFG_Contraception_guidance_Version_1.1.pdf)
* Hypersensitivity to the active ingredient or any excipients of the investigational drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-11-21 (Estimated); Study Completion 2027-03-21 (Estimated)

PRIMARY OUTCOMES:
Emergent Adverse Events assessed by physical and neurological examination | Clinical follow-up every month for 2 years
  Information on adverse events will be reviewed through direct questioning of the patient.
Emergent Adverse Events assessed by evaluation of the results of the analysis with hematology and biochemistry. | Clinical follow-up every month for 2 years
  Information on adverse events will be reviewed through the results of examinations, complementary tests and analytical parameters.
Emergent Adverse Events assessed by brain RM image | every 3 months after surgery, for 2 years
  brain RM image, for neuroradiological follow-up
Emergent Adverse Events assessed by AC_PET with 18-FdG | every 6 months after surgery, for 2 years
  AC_PET image, for neuroradiological follow-up

SECONDARY OUTCOMES:
Efficacy assessed by progression-free survival (PFS) | through study completion, an average of 2 yeas.
  Progression-free survival (PFS), a measure of how long a patient receives treatment before the cancer begins to grow.
Efficacy assessed by overall survival (OS) | through study completion, an average of 2 yeas.
  Overall survival (OS), how long patients live after starting treatment.
Quality of life assessed by The Functional Assessment of Cancer Therapy-Brain (FACT-Br) | every 3 months after surgery, for 2 years
  A commonly used instrument measuring general quality of life (QOL) that reflects symptoms or problems associated with brain malignancies across 5 scales. Patients rate all 5 items using a five-point Likert scale ranging from 0 "not at all" to 4 "very much." Overall, higher ratings suggest higher QOL
Cognitive functionality assessed by MONTREAL COGNITIVE ASSESSMENT (MOCA) | every 3 months after surgery, for 2 years
  It has been shown to be useful at detecting cognitive dysfunction in brain metastases.
  The test is a one-page, 30-point test that can be administered in 10 minutes. It assesses short-term memory recall (5 points), visuospatial abilities through clock-drawing (3 points) and cube copy (1 point), and orientation (6 points). Executive function is assessed through modified Trail Making Part B (1 point), phonemic fluency (1 point), and verbal abstraction (2 points). A sustained-attention task (1 point), digit span (2 points), and serial calculation (3 points) test attention, concentration, and working memory. And lastly, language is assessed through naming low-familiarity animals (3 points), sentence repetition (2 points), and the fluency task

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain